CLINICAL TRIAL: NCT02294682
Title: A Phase II, Randomized, Multicenter, Dose-Ranging Study in Adult Subjects Evaluating the Efficacy, Safety, and Tolerability of Single Doses of GSK2140944 in the Treatment of Uncomplicated Urogenital Gonorrhea Caused by Neisseria Gonorrhoeae
Brief Title: A Dose-Ranging Study Evaluating the Efficacy, Safety, and Tolerability of GSK2140944 in the Treatment of Uncomplicated Urogenital Gonorrhea Caused by Neisseria Gonorrhoeae
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116576
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-02

CONDITIONS: Gonorrhea
Keywords: uncomplicated urogenital gonorrhea; Bacterial Type II Topoisomerase Inhibitors (BTI); antibiotics; GSK2140944; N. gonorrhoeae
MeSH Terms: conditions — Gonorrhea | interventions — gepotidacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2140944 1500 mg (Experimental): Subjects will receive single oral dose of GSK2140944 1500 mg.
  Interventions: Drug: GSK2140944
- GSK2140944 3000 mg (Experimental): Subjects will receive single oral dose of GSK2140944 3000 mg.
  Interventions: Drug: GSK2140944

INTERVENTIONS:
Drug: GSK2140944 — Immediate release capsules (pink hard gelatin size 00 capsule, with no external marking, filled with slightly agglomerated pale yellowish to grayish yellow powder) containing GSK2140944 500 mg and inactive formulation excipients. GSK2140944 will be administered orally once 1500 mg (3 capsules) or 3000 mg (6 capsules).

SUMMARY:
GSK2140944 has demonstrated in vitro activity against Neisseria (N.) gonorrhoeae, including ciprofloxacin resistant and susceptible strains. This study is a Phase II, randomized, multicenter, open-label, dose ranging study designed to inform the optimal oral dose of GSK2140944 by further characterizing the efficacy, safety, and tolerability in subjects with uncomplicated urogenital gonorrhea due to N. gonorrhoeae. Subjects will be randomly assigned to receive either a single 1500 milligrams (mg) or 3000 mg oral dose of GSK2140944. Appropriate safety and microbiological assessments will be conducted at the Baseline (Day 1) Visit and repeated at the Test-of-Cure (Day 4 to 8) Visit. The study duration will be approximately 1 week. Approximately 60 microbiologically evaluable subjects (30 subjects in each treatment arm) will complete the study if both arms remain active throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adult male or female at least 18 years of age at the time of signing informed consent who meets one of the following criteria:

  1. A non-pregnant, non-lactating female of childbearing potential who 1) is sexually inactive by abstinence, 2) has a sole male partner who has been sterilized, or 3) uses a contraceptive method with a failure rate of <1% through the Test-of-Cure Visit. Females of childbearing potential must not become pregnant during the study.
  2. A female of non-childbearing potential, which includes the following: Females who are surgically sterile with a documented hysterectomy and/or bilateral oophorectomy; Females with documented tubal ligation. If the procedure was done hysteroscopically, the effectiveness of tubal occlusion must have been documented by hysterosalpingogram after the procedure (typically 3 months after the procedure); Females who are post-menopausal, defined as amenorrhoeic for greater than 1 year. For women whose menopausal status is in doubt, documented previous confirmatory blood samples with follicle-stimulating hormone >40 milli international units (mIU)/millilitre (mL) and estradiol <40 picograms (pg)/mL (<140 picomoles [pmol]/litre [L]) will need to be confirmed, or they will be required to use one of the acceptable contraception methods. Note: For the purposes of these criteria, "documented" includes information obtained via a verbal interview with the subject or from the subject's medical records.
* There is clinical suspicion that the subject has a urogenital gonococcal infection (e.g., prior culture, nucleic acid amplification test [NAAT] or Gram stain presumptive or positive for the presence of N. gonorrhoeae, or sexual contact with a partner diagnosed with gonorrhea within the past 14 days, as reported by the subject). Note: All subjects will be tested for N. gonorrhoeae, but these results will not be used to determine subject eligibility for enrollment in the study.
* The subject has provided written, dated, informed consent and is willing and able to comply with the study protocol.

Exclusion Criteria:

* The subject is pregnant or nursing.
* The subject is a hysterectomized female without a cervix.
* The subject is a male with a current diagnosis of epididymitis or orchitis at the time of the Baseline Visit.
* The subject has a body mass index >=40.0 kilograms (kg)/square meter (m^2).
* The subject has a serious underlying disease that could be imminently life threatening, or the subject is unlikely to survive for the duration of the study period.
* The subject has a medical condition or requires medication that may be aggravated by inhibition of acetylcholinesterase, such as: Poorly controlled asthma or chronic obstructive pulmonary disease at baseline and, in the opinion of the investigator, is not stable on current therapy; Acute severe pain, uncontrolled with conventional medical management; Active peptic ulcer disease; Parkinson's disease; Myasthenia gravis; A history of seizure disorder requiring medications for control. This does not include a history of childhood febrile seizures; Any evidence of mechanical obstruction of the urinary or digestive tracks.
* The subject has had any past history or current diagnosis of Clostridium difficile infection at the time of the Baseline Visit.
* The subject, in the judgment of the investigator, would not be able or willing to comply with the protocol or complete study follow-up.
* The subject has a history of sensitivity to the study medication, or components thereof, or a history of a drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* The subject has a PR interval <120 or >220 milliseconds (msec). Note: Subjects without an evaluable PR interval (e.g., stable atrial fibrillation) are not eligible for this study.
* The subject has a corrected QT (QTc) >450 msec or a QTc >480 msec for subjects with bundle branch block. Note: The QTc is the QT interval corrected for heart rate according to either Bazett formula (QTcB), Fridericia formula (QTcF), machine, or manual overread.
* The subject has QRS duration <70 or >120 msec.
* The subject has pre-existing Grade II atrioventricular block or higher or a history of significant vasovagal and/or syncopal episodes or episodes of symptomatic bradycardia.
* The subject has a current or chronic history of liver disease (with the exception of Gilbert's syndrome), including symptomatic viral hepatitis and moderate to severe liver insufficiency (Child Pugh class B or C).
* The subject has been previously enrolled in this study or has previously been treated with GSK2140944.
* The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer.
* The subject has the following gonococcal infections: Suspected or confirmed pelvic inflammatory disease; Suspected or confirmed gonococcal arthritis; Other evidence of disseminated gonococcal infection.
* The subject has received treatment with a systemic or intravaginal antibacterial within 14 days of study entry.
* Subject is taking a medication that has a known risk of torsades de pointes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-04-15; Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (11):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Jenkintown, Pennsylvania
- GSK Investigational Site, San Juan, Puerto Rico
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Scangarella-Oman NE, Hossain M, Perry CR, Tiffany C, Powell M, Swift B, Dumont EF. Dose selection for a phase III study evaluating gepotidacin (GSK2140944) in the treatment of uncomplicated urogenital gonorrhoea. Sex Transm Infect. 2023 Feb;99(1):64-69. doi: 10.1136/sextrans-2022-055518. Epub 2022 Nov 21. PMID 36411033
- [Derived] Scangarella-Oman NE, Hossain M, Dixon PB, Ingraham K, Min S, Tiffany CA, Perry CR, Raychaudhuri A, Dumont EF, Huang J, Hook EW 3rd, Miller LA. Microbiological Analysis from a Phase 2 Randomized Study in Adults Evaluating Single Oral Doses of Gepotidacin in the Treatment of Uncomplicated Urogenital Gonorrhea Caused by Neisseria gonorrhoeae. Antimicrob Agents Chemother. 2018 Nov 26;62(12):e01221-18. doi: 10.1128/AAC.01221-18. Print 2018 Dec. PMID 30249694
- [Derived] Taylor SN, Morris DH, Avery AK, Workowski KA, Batteiger BE, Tiffany CA, Perry CR, Raychaudhuri A, Scangarella-Oman NE, Hossain M, Dumont EF. Gepotidacin for the Treatment of Uncomplicated Urogenital Gonorrhea: A Phase 2, Randomized, Dose-Ranging, Single-Oral Dose Evaluation. Clin Infect Dis. 2018 Aug 1;67(4):504-512. doi: 10.1093/cid/ciy145. PMID 29617982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase II, randomized, multicenter, open-label, dose ranging study evaluating the efficacy, safety and tolerability of gepotidacin therapy in participants with uncomplicated urogenital gonorrhea. The study duration was approximately 1 week with 2 planned study visits: Baseline (Day 1, pre-dose) and Test-of-Cure (TOC) (Day 4 to 8) visit.
Pre-assignment Details: A total of 106 participants (par.) were randomized to receive GSK2140944 1500 milligrams (mg) or GSK2140944 3000 mg, of which 105 participants received any dose of study treatment and 1 par. was unable to swallow the capsule; therefore, did not receive study drug.
Groups:
- GSK2140944 1500 mg: Participants were randomized to receive oral dose of GSK2140944 1500 mg (3 immediate-release capsules of 500 mg each) with food and 240 milliliters (mL) of water. Additional 100 mL of water was given to assist in swallowing a large number of capsules. Participants who tested positive for chlamydia trachomatis at the Baseline visit, received a single 1 gram dose of azithromycin or local standard of care at the TOC visit.
- GSK2140944 3000 mg: Participants were randomized to receive oral dose of GSK2140944 3000 mg (6 immediate-release capsules of 500 mg each) with food and 240 mL of water. Additional 100 mL of water was given to assist in swallowing a large number of capsules. Participants who tested positive for chlamydia trachomatis at the Baseline visit, received a single 1 gram dose of azithromycin or local standard of care at the TOC visit.
Period: Overall Study
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Started | 53 | 53
Completed | 52 | 53
Not Completed | 1 | 0
Not completed — Could not swallow pills | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (11.45) | 32.4 (11.33) | 33.3 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 50 | 51 | 101
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage (Heri.) | 22 | 25 | 47
  American Indian or Alaska Native | 1 | 1 | 2
  Central/South Asian Heritage | 0 | 1 | 1
  Japanese/East Asian Heri. /South East Asian Heri. | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 24 | 21 | 45
  White & African American/African Heritage | 0 | 1 | 1
  Unknown | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Culture-confirmed Bacterial Eradication of Urogenital Neisseria Gonorrhoeae at the Test-of-Cure Visit
Description: Pre-treatment urogenital, pharyngeal, and rectal swab specimens were obtained for bacteriological culture for neisseria (N.) gonorrhoeae at the Baseline visit. Test- of-Cure was defined by infection site (that is urogenital and, as appropriate, rectal and/or pharyngeal) as culture confirmed bacterial eradication of N. gonorrhoeae observed 3 to 7 days post-treatment. Pre-treatment urogenital specimens were obtained for nucleic acid amplification test (NAAT) assay to detect the presence of N. gonorrhoeae and chlamydia trachomatis at the Baseline visit. Only participants who had a pre-therapy N. gonorrhoeae isolate recovered from their urogenital specimen were evaluated. Microbiologically evaluable (ME) Population comprised of all randomized participants who had N. gonorrhoeae isolated from Baseline cultures of urogenital swab specimens, received any dose of gepotidacin, and returned for their TOC visit.
Time Frame: Baseline (Day 1, pre-dose) and Test-of-Cure visit (Day 4 to 8)
Population: ME Population
Measure: Number; unit: Participants
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 30 | 39
Participants | 29 | 37
Statistical Analysis 1: Comparison: GSK2140944 1500 mg; Test type: Superiority or Other; Microbio Response Urogenital Gonorrhea = 97, 95% CI 1-sided [lower limit 85.1] — GSK2140944 1500 mg
Statistical Analysis 2: Comparison: GSK2140944 3000 mg; Test type: Superiority or Other; Microbio Response Urogenital Gonorrhea = 95, 95% CI 1-sided [lower limit 84.7] — GSK2140944 3000 mg

2. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participants, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinaemia (defined as alanine aminotransferase [ALT] >=3 times upper limit of normal [ULN] and bilirubin >=2 times ULN [>35 percent direct] [or ALT >=3 times ULN and international normalization ratio INR>1.5, if INR is measured].
Time Frame: From start of the study treatment until Test-of-Cure visit (Day 4 to 8)
Population: Safety Population: comprised of all randomized participants who received any dose of study medication.
Measure: Number; unit: Participants
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Participants
  Any AE | 27 | 34
  Any SAE | 0 | 0

3. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at the Indicated Time Points
Description: BP was measured in semi-supine position after 5 minutes rest. It was recorded at Baseline visit, 2 hour post-dose visit for participants enrolled under orignal protocol, 0.5 hour post-dose for participants enrolled under protocol amendement 1 and up to TOC visit (Day 4 to 8).Vital sign measurements were obtained prior to any scheduled blood collection visit on the same assessment day. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as TOC visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit (Day 1) and Day 4 to Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Millimeter of mercury (mmHg)
  Systolic BP, Day 1, 2 hr post-dose, n=47, 48 | 0.4 (11.61) | 1.3 (11.97)
  Systolic BP, Day 4 to 8, n=52, 53 | -2.8 (13.11) | 0.5 (11.73)
  Diastolic BP, Day 1, 2 hr post-dose, n=47, 48 | 0.1 (7.61) | -0.9 (8.40)
  Diastolic BP, Day 4 to 8, n=52, 53 | -2.3 (8.73) | -2.2 (9.86)

4. Secondary Outcome: Change From Baseline in Pulse Rate at the Indicated Time Points
Description: Pulse rate was measured in semi-supine position after 5 minutes rest. It was recorded at Baseline visit, 2 hour post-dose visit for participants enrolled under orignal protocol, 0.5 hour post-dose for participants enrolled under protocol amendement 1 and up to TOC visit (Day 4 to 8). Vital sign measurements were obtained prior to any scheduled blood collection visit on the same assessment day. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as TOC visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit (Day 1) and Day 4 to Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Beats per minute
  Pulse rate Day 1, 2 hr post-dose, n=47, 48 | -0.3 (12.20) | -1.4 (8.72)
  Pulse rate, Day 4 to 8, n=52, 53 | 1.1 (11.92) | 2.2 (14.12)

5. Secondary Outcome: Change From Baseline in Temperature at the Indicated Time Points
Description: Temperature was measured in semi-supine position after 5 minutes rest. It was recorded at Baseline visit, 2 hour post-dose visit for participants enrolled under orignal protocol, 0.5 hour post-dose for participants enrolled under protocol amendement 1 and up to TOC visit (Day 4 to 8). Vital sign measurements were obtained prior to any scheduled blood collection visit on the same assessment day. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as TOC visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit (Day 1) and Day 4 to Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Celsius
  Temperature, Day 1, 2 hr post-dose, n=47, 48 | -0.126 (0.4327) | -0.052 (0.3664)
  Temperature, Day 4 to 8, n=52, 53 | -0.121 (0.4953) | -0.088 (0.3742)

6. Secondary Outcome: Change From Baseline in Respiratory Rate at the Indicated Time Points
Description: Respiratory rate was measured in semi-supine position after 5 minutes rest. It was recorded at Baseline visit, 2 hour post-dose visit for participants enrolled under orignal protocol, 0.5 hour post-dose for participants enrolled under protocol amendement 1 and up to TOC visit (Day 4 to 8). Vital sign measurements was obtained prior to any scheduled blood collection visit on the same assessment day. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as TOC Visit value minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit (Day 1) and Day 4 to Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Breaths per minute
  Respiratory rate, Day 1, 2 hr post-dose, n=47, 48 | -0.1 (1.39) | -0.3 (1.51)
  Respiratory rate, Day 4 to 8, n=52, 53 | 0.1 (1.66) | -0.1 (1.61)

7. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: A single 12-lead ECGs were obtained at the Baseline, 2 hour post-dose, and at the TOC (Day 4 to 8) visit using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals. ECG was obtained prior to any vital sign measurements or blood draws scheduled on the same assessment day. For participants enrolled under protocol amendment 1, ECG was measured at Baseline visit Day 1 (pre-dose) only. ECG assessments were presented as abnormal-clinically significant (CS) and abnormal-not clinically significant (NCS) at the indicated time points. Only those participants available at the specified time points were analyzed (represented by n=X , X in the category titles).
Time Frame: Baseline visit and up to Day 8
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Participants
  Abnormal-NCS, pre-dose Day 1, n=52, 53 | 14 | 12
  Abnormal-CS, pre-dose Day 1, n=52, 53 | 0 | 0
  Abnormal-NCS, Day 1, 2 hr post, n=37, 36 | 8 | 9
  Abnormal-CS, Day 1, 2 hr post, n=37, 36 | 0 | 0
  Abnormal-NCS, Day 4 to 8, n=37, 35 | 7 | 11
  Abnormal-CS, Day 4 to 8, n=37, 35 | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Physical Examination Finding
Description: Physical examination of respiratory, cardiovascular, abdomen, gastrointestinal, urogenital systems, pharyngeal and rectal examinations with collections of microbiology specimen was performed at the Baseline and TOC (Day 4 to 8) visit. Baseline was defined as the study assessment on Day 1 (pre-dose). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Participants
  Abdomen, Baseline, n=50, 53 | 2 | 0
  Abdomen, TOC, n=51, 52 | 0 | 0
  Cardiovascular, Baseline, n=52, 53 | 1 | 1
  Cardiovascular, TOC, n=51, 53 | 0 | 0
  Gastrointestinal, Baseline, n=49, 52 | 1 | 0
  Gastrointestinal, TOC, n=50, 51 | 2 | 0
  Pharyngeal, Baseline, n=51, 51 | 1 | 4
  Pharyngeal, TOC, n=51, 52 | 0 | 0
  Rectal examination, Baseline, n=46, 46 | 2 | 4
  Rectal examination, TOC, n=41, 42 | 1 | 2
  Respiratory, Baseline, n=52, 53 | 1 | 0
  Respiratory, TOC, n=52, 53 | 0 | 0
  Urogenital, Baseline, n=52, 53 | 49 | 47
  Urogenital, TOC, n=52, 51 | 5 | 6

9. Secondary Outcome: Change From Baseline in Hemoglobin, Protein and Albumin at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1 (pre-dose) and at TOC visit (Day 4 to 8) to evaluate hemoglobin, total protein and albumin. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Gram (G)/Liter (L)
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Gram (G)/Liter (L)
  Hemoglobin, n=46, 53 | -3.0 (6.89) | -3.9 (8.79)
  Albumin, n=52, 53 | -0.5 (2.10) | -0.8 (2.51)
  Protein, n=52, 53 | -1.1 (3.62) | -2.0 (4.01)

10. Secondary Outcome: Change From Baseline in Hematocrit at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1 (pre-dose) and at TOC visit (Day 4 to 8) to evaluate hematocrit. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of blood
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 46 | 53
Proportion of blood | -0.0117 (0.02213) | -0.0155 (0.03166)

11. Secondary Outcome: Change From Baseline in Lymphocyte, Monocyte, Neutrophil Basophil, Eosinophil, Leukocyte and Platelet Count at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1 (pre-dose) and at TOC visit (Day 4 to 8) to evaluate neutrophil, lymphocyte, basophil, eosinophil, monocyte, leukocyte and platelet count. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
10^9 cells/L
  Lymphocytes, n=46, 52 | 0.141 (0.5437) | 0.053 (0.6846)
  Monocytes, n=46, 52 | -0.013 (0.1339) | 0.026 (0.1377)
  Neutrophils , n=46, 52 | -0.834 (1.7564) | -0.598 (1.9185)
  Platelets, n=45, 53 | 6.4 (35.63) | -5.8 (26.41)
  Basophils, n=46, 52 | -0.001 (0.0146) | 0.002 (0.0155)
  Eosinophils, n=46, 52 | 0.023 (0.1147) | 0.027 (0.1187)
  Leukocytes, n=46, 52 | -0.69 (1.692) | -0.49 (1.947)

12. Secondary Outcome: Change From Baseline in Bilirubin, Direct Bilirubin and Creatinine at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1 (pre-dose) and at TOC visit (Day 4 to 8) to evaluate bilirubin, direct bilirubin and creatinine. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromole (UMOL)/ L
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Micromole (UMOL)/ L
  Bilirubin, n=52, 53 | -1.4 (5.42) | 0.4 (4.01)
  Direct bilirubin, n=52, 53 | -0.2 (1.11) | 0.2 (1.45)
  Creatinine, n=52, 53 | 1.38 (9.989) | 2.01 (7.737)

13. Secondary Outcome: Change From Baseline in Alanine Aminotransferase, Aspartate Aminotransferase and Alkaline Phosphatase at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1.(pre-dose) and at TOC visit (Day 4 to 8) to evaluate alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units (IU)/ L
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
International units (IU)/ L
  Alanine Aminotransferase, n=52, 53 | 1.2 (7.24) | 1.8 (8.41)
  Aspartate Aminotransferase, n=52, 53 | 2.0 (7.69) | 2.5 (8.69)
  Alkaline Phosphatase, n=52, 53 | -1.8 (6.73) | -2.2 (6.26)

14. Secondary Outcome: Change From Baseline in Chloride, Calcium, Glucose, Potassium, Sodium and Urea at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1.(pre-dose) and at TOC visit (Day 4 to 8) to evaluate chloride, calcium, glucose, potassium, sodium and urea (blood urea nitrogen). Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimole (MMOL)/L
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Millimole (MMOL)/L
  Chloride, n=52, 53 | 0.7 (2.02) | 0.3 (1.92)
  Calcium, n=52, 53 | -0.017 (0.0869) | -0.047 (0.0874)
  Glucose, n=52, 53 | -0.18 (1.184) | -0.02 (0.959)
  Potassium, n=52, 53 | 0.04 (0.359) | -0.01 (0.355)
  Sodium, n=52, 53 | 0.1 (2.28) | -0.1 (1.95)
  Urea, n=52, 53 | 0.07 (1.098) | 0.04 (1.228)

15. Secondary Outcome: Change From Baseline in Erythrocytes at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1 (pre-dose) and at TOC visit (Day 4 to 8) to evaluate erythrocytes (red blood cell count). Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 46 | 53
10^12/L | -0.10 (0.227) | -0.15 (0.338)

16. Secondary Outcome: Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1 (pre-dose) and at TOC visit (Day 4 to 8) to evaluate erythrocytes mean corpuscular hemoglobin. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC Visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 46 | 53
Picograms | 0.08 (0.457) | 0.12 (0.461)

17. Secondary Outcome: Change From Baseline in Erythrocytes Mean Corpuscular Volume at Test-of-Cure Visit (Day 4 to 8)
Description: Blood samples were collected at Baseline Day 1 (pre-dose) and at TOC visit (Day 4 to 8) to evaluate erythrocytes mean corpuscular volume. Baseline was defined as the study assessment on Day 1 (pre-dose). Change from Baseline was calculated as value obtained at TOC Visit minus value at Baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 46 | 53
Femtoliters | -0.3 (1.85) | -0.2 (1.71)

18. Secondary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results
Description: Dipstick urinalysis was done for glucose, ketones, occult blood, protein, potential hydrogen (pH) and specific gravity at Baseline visit Day 1 (pre-dose) and Test-of-Cure visit (Day 4 to 8). Results were presented as negative (normal) or other findings reported only if observed under microscopic examination trace, 1+, 2+, 3+, 4+ and 5+ glucose, ketones, occult blood and protein. pH results were categorized as per their pH values. Baseline was defined as the study assessment on Day 1 (pre-dose). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline visit and Test-of-Cure visit (Day 4 to 8)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Number analyzed (Participants) | 52 | 53
Participants
  Glucose, pre-dose, Day 1, negative, n=50, 53 | 48 | 53
  Glucose, pre-dose, Day 1, trace, n=50, 53 | 1 | 0
  Glucose, pre-dose, Day 1, 1+, n=50, 53 | 0 | 0
  Glucose, pre-dose, Day 1, 2+, n=50, 53 | 0 | 0
  Glucose, pre-dose, Day 1, 3+, n=50, 53 | 1 | 0
  Glucose, pre-dose, Day 1, 4+, n=50, 53 | 0 | 0
  Glucose, pre-dose, Day 1, 5+, n=50, 53 | 0 | 0
  Glucose, Day 4 to 8, negative, n=48, 53 | 47 | 53
  Glucose, Day 4 to 8, trace, n=48, 53 | 0 | 0
  Glucose, Day 4 to 8, 1+, n=48, 53 | 0 | 0
  Glucose, Day 4 to 8, 2+, n=48, 53 | 0 | 0
  Glucose, Day 4 to 8, 3+, n=48, 53 | 1 | 0
  Glucose, Day 4 to 8, 4+, n=48, 53 | 0 | 0
  Glucose, Day 4 to 8, 5+, n=48, 53 | 0 | 0
  Ketones, pre-dose, Day 1, negative, n=50, 53 | 48 | 49
  Ketones, pre-dose, Day 1, trace, n=50, 53 | 2 | 3
  Ketones, pre-dose, Day 1, 1+, n=50, 53 | 0 | 1
  Ketones, pre-dose, Day 1, 2+, n=50, 53 | 0 | 0
  Ketones, pre-dose, Day 1, 3+, n=50, 53 | 0 | 0
  Ketones, pre-dose, Day 1, 4+, n=50, 53 | 0 | 0
  Ketones, pre-dose, Day 1, 5+, n=50, 53 | 0 | 0
  Ketones, Day 4 to 8, negative, n=48, 53 | 45 | 48
  Ketones, Day 4 to 8, trace, n=48, 53 | 3 | 4
  Ketones, Day 4 to 8, 1+, n=48, 53 | 0 | 1
  Ketones, Day 4 to 8, 2+, n=48, 53 | 0 | 0
  Ketones, Day 4 to 8, 3+, n=48, 53 | 0 | 0
  Ketones, Day 4 to 8, 4+, n=48, 53 | 0 | 0
  Ketones, Day 4 to 8, 5+, n=48, 53 | 0 | 0
  Occult blood, pre-dose, Day 1, negative, n=50, 53 | 35 | 42
  Occult blood, pre-dose, Day 1, trace, n=50, 53 | 6 | 4
  Occult blood, pre-dose, Day 1, 1+, n=50, 53 | 6 | 7
  Occult blood, pre-dose, Day 1, 2+, n=50, 53 | 2 | 0
  Occult blood, pre-dose, Day 1, 3+, n=50, 53 | 1 | 0
  Occult blood, pre-dose, Day 1, 4+, n=50, 53 | 0 | 0
  Occult blood, pre-dose, Day 1, 5+, n=50, 53 | 0 | 0
  Occult blood, Day 4 to 8, negative, n=48, 53 | 45 | 49
  Occult blood, Day 4 to 8, trace, n=48, 53 | 0 | 0
  Occult blood, Day 4 to 8, 1+, n=48, 53 | 1 | 1
  Occult blood, Day 4 to 8, 2+, n=48, 53 | 2 | 0
  Occult blood, Day 4 to 8, 3+, n=48, 53 | 0 | 3
  Occult blood, Day 4 to 8, 4+, n=48, 53 | 0 | 0
  Occult blood, Day 4 to 8, 5+, n=48, 53 | 0 | 0
  Protein, pre-dose, Day 1, negative, n=50, 53 | 37 | 39
  Protein, pre-dose, Day 1, trace, n=50, 53 | 8 | 9
  Protein, pre-dose, Day 1, 1+, n=50, 53 | 4 | 5
  Protein, pre-dose, Day 1, 2+, n=50, 53 | 1 | 0
  Protein, pre-dose, Day 1, 3+, n=50, 53 | 0 | 0
  Protein, pre-dose, Day 1, 4+, n=50, 53 | 0 | 0
  Protein, pre-dose, Day 1, 5+, n=50, 53 | 0 | 0
  Protein, Day 4 to 8, negative, n=48, 53 | 42 | 43
  Protein, Day 4 to 8, trace, n=48, 53 | 4 | 7
  Protein, Day 4 to 8, 1+, n=48, 53 | 2 | 2
  Protein, Day 4 to 8, 2+, n=48, 53 | 0 | 1
  Protein, Day 4 to 8, 3+, n=48, 53 | 0 | 0
  Protein, Day 4 to 8, 4+, n=48, 53 | 0 | 0
  Protein, Day 4 to 8, 5+, n=48, 53 | 0 | 0
  pH, pre-dose, Day 1, pH 5, n=50, 53 | 2 | 1
  pH, pre-dose, Day 1, pH 5.5, n=50, 53 | 5 | 8
  pH, pre-dose, Day 1, pH 6, n=50, 53 | 13 | 8
  pH, pre-dose, Day 1, pH 6.5, n=50, 53 | 12 | 14
  pH, pre-dose, Day 1, pH 7, n=50, 53 | 12 | 14
  pH, pre-dose, Day 1,pH 7.5 ,n=50, 53 | 4 | 7
  pH, pre-dose, Day 1, pH 8, n=50, 53 | 2 | 1
  pH, Day 4 to 8, pH 5, n=48, 53 | 0 | 0
  pH, Day 4 to 8, pH 5.5, n=48, 53 | 10 | 11
  pH, Day 4 to 8, pH 6, n=48, 53 | 13 | 15
  pH, Day 4 to 8, pH 6.5, n=48, 53 | 9 | 14
  pH, Day 4 to 8, pH 7, n=48, 53 | 10 | 7
  pH, Day 4 to 8, pH 7.5, n=48, 53 | 5 | 3
  pH, Day 4 to 8, pH 8, n=48, 53 | 1 | 3

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of the study treatment (Day1) until Test-of-Cure visit (Day 4 to 8).
Description: On-treatment SAEs and non-serious (AEs) are reported for Safety Population which comprised of all randomized participants who received any dose of study medication.
Arm/Group | GSK2140944 1500 mg | GSK2140944 3000 mg
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 22/52 | 28/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2140944 1500 mg (N=52) | GSK2140944 3000 mg (N=53)
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 9 | 19
Eructation (Gastrointestinal disorders) | 1 | 3
Faeces soft (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 14 | 10
Nausea (Gastrointestinal disorders) | 3 | 11
Fatigue (General disorders) | 3 | 5
Feeling hot (General disorders) | 1 | 4
Dizziness (Nervous system disorders) | 1 | 6
Somnolence (Nervous system disorders) | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.